CLINICAL TRIAL: NCT05135845
Title: Phase II Trial to Evaluate the Combination of Capmatinib + Spartalizumab in Advanced Oesogastric Adenocarcinoma
Brief Title: Combination of Capmatinib + Spartalizumab in Advanced Oesogastric Adenocarcinoma
Acronym: METIMGAST
Status: Suspended | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor decision up DSMB advice due to unfavorable toxicity profile
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APHP201152
Record Dates: First submitted 2021-10-28; First posted 2021-11-26 (Actual); Last update posted 2023-02-03 (Actual); Status verified 2023-01

CONDITIONS: Oesophageal Adenocarcinoma; Gastric Adenocarcinoma
MeSH Terms: conditions — Adenocarcinoma Of Esophagus | interventions — capmatinib; spartalizumab

STUDY DESIGN:
Intervention Model Description: Multicenter single-arm adaptive phase II trial with 2 cohorts according to MET amplification level :
  * Cohort 1: tumor without MET amplification (< 6 copies);
  * Cohort 2: tumor with MET amplification (≥6 copies).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Capmatinib — Capmatinib 400mg BID for a maximum of 12 months or until progression, patient's refusal or unacceptable toxicity
  Other Names: INC280
Drug: Spartalizumab — Spartalizumab 300mg Q3W for a maximum of 12 months or until progression, patient's refusal or unacceptable toxicity
  Other Names: PDR001

SUMMARY:
Immunotherapy with anti-PD1 antibodies provides encouraging results on a subset of patients. Capmatinib, a MET inhibitor, has shown an imunomodulatory effect and a synergy with spartalizumab a PD-1 inhibitor. The purpose of this phase II trial is to evaluate the efficacy and safety of the combination of capmatinib + spartalizumab in adult patients with advanced oesogastric adenocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically documented locally advanced or metastatic oesogastric adenocarcinoma.
* Unresectable tumor.
* Patients must have received at least one prior systemic chemotherapy based on platinium salt and fluoropyrimidine with documented progression during chemotherapy.
* Patients must have received trastuzumab in case of HER2 positive tumor (HER2 +++ or HER2++ and FISH or SISH+)
* Determination of tumor MET amplification by FISH available
* ECOG Performance Status ≤ 1.
* Measurable tumoral disease according to RECIST 1.1 criteria.
* Patients must be willing and able to swallow and retain oral medication.
* Age ≥18 years.
* Women of childbearing potential and males who are sexually active must agree to follow instructions for method(s) of contraception for the duration of study treatments with Capmatinib and Spartalizumab until 7 days after the last dose of Capmatinib and 150 days after the last dose of Spartalizumab
* Consent to participate in the trial after information
* Affiliated to a social security system

Exclusion Criteria:

* Previous treatment with immunotherapy or MET inhibitor
* Impossibility to take oral medication
* Persistent toxicities related to prior treatment of grade greater than 1
* Presence or history of another malignant disease that has been diagnosed and/or required therapy within the past 3 years. Exceptions to this exclusion include: completely resected basal cell and squamous cell skin cancers, and completely resected carcinoma in situ of any type.
* Use of any live vaccines within 4 weeks of initiation of study treatment.
* History of severe hypersensitivity reactions to other monoclonal antibodies (mAbs).
* History or current interstitial lung disease or non-infectious pneumonitis
* Active autoimmune disease or a documented history of autoimmune disease (Patients with vitiligo, controlled type I diabetes mellitus on stable insulin dose, residual autoimmune-related hypothyroidism only requiring hormone replacement or psoriasis not requiring systemic treatment are permitted).
* Allogenic bone marrow or solid organ transplant
* Uncontrolled active infection
* Human Immunodeficiency Virus (HIV) infection
* Untreated active Hepatitis B infection (HBsAg positive) (Patients with active hepatitis B (HBsAg positive) may be enrolled provided viral load (HBV DNA) at screening is <100 UI/mL. Patients may receive antiviral treatment with lamivudine, tenofovir, entecavir, or other antiviral agents before the initiation of study treatment to suppress viral replication).
* Untreated active hepatitis C (HCV RNA positive) (patients that achieved a sustained virological response after antiviral treatment and show absence of detectable HCV RNA ≥6 months after cessation of antiviral treatment are eligible)
* Untreated or symptomatic central nervous system (CNS) lesion. However, patients are eligible if: a) all known CNS lesions have been treated with radiotherapy or surgery and b) patient remained without evidence of CNS disease progression ≥4 weeks after treatment and c) patients must be off corticosteroid therapy for ≥2 weeks
* Clinically significant, uncontrolled heart diseases
* Recent acute coronary syndrome or unstable ischemic heart disease
* Congestive heart failure ≥ Class III or IV as defined by New York Heart Association
* Long QT syndrome (> 480 ms in women and 470 ms in men), family history of idiopathic sudden death or congenital long QT syndrome.
* Uncontrolled hypertension defined by a Systolic Blood Pressure (SBP) ≥150 mm Hg and/or Diastolic Blood Pressure (DBP) ≥ 100 mm Hg, with or without antihypertensive medication. Initiation or adjustment of antihypertensive medication(s) is allowed prior to screening
* Surgery less than 4 weeks
* Radiotherapy less than 2 weeks
* Pregnancy or breastfeeding or women of child-bearing potential, unless they are using highly effective methods of contraception.
* Sexually active males unless they use a condom during intercourse while taking capmatinib and for 7 days after stopping treatment and should not father a child in this period.
* Participants receiving treatment with strong inducers of CYP3A and could not be discontinued ≥ 1 week prior to the start of treatment.
* Systemic chronic steroid therapy (>10 mg/day prednisone or equivalent) or any immunosuppressive therapy 7 days prior to planned date of first dose of study treatment.
* Patient having out of range laboratory values defined as:
* Total bilirubin >2 mg/dL, except for patients with Gilbert's syndrome who are excluded if total bilirubin >3.0 x ULN or direct bilirubin >1.5 x ULN
* Alanine aminotransferase (ALT) > 3 x ULN
* Aspartate aminotransferase (AST) > 3 x ULN
* Coagulation: Prothrombin Time (PT) >4 seconds more than the ULN or International Normalized Ratio (INR) >1.7
* Absolute neutrophil count (ANC) <1.5 x 109/L
* Platelet count <75 x 109/L
* Hemoglobin <9 g/dL
* Creatinine clearance (calculated using Cockcroft-Gault formula, or measured) <45 mL/min
* Serum lipase >1 ULN
* Cardiac troponin I (cTnI) elevation >2 x ULN
* Potassium, Magnesium, Phosphorus, total Calcium (corrected for serum albumin) outside of normal limits (patients may be enrolled if corrected to within normal limits with supplements during screening)
* Patients under legal protection
* Participation to another interventional study with treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2022-03-22 (Actual); Primary Completion 2023-04 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Tumor response | 6 months
  Overall response rate defined as the proportion of patients with at least one objective tumour response (complete or partial) according to response evaluation criteria in solid tumours (RECIST) v1.1 within 6 months.

SECONDARY OUTCOMES:
Proportion of unacceptable toxicity of the regimen during the first and second cycles of administration | Day 42
  Presence of at least one of (composite endpoint):
  * Adverse event (AE) grade >3 (NCI-CTCAE v5), at least possibly related to the treatment or unrelated to disease, progression, intercurrent illness, concomitant medications
  * Non-hematological AE grade ≥3
  * Recurring grade 2 pneumonitis, Myocarditis grade ≥2
  * Autoimmune hemolytic anemia, hemolytic uremic syndrome, acquired hemophilia grade ≥3
  * Guillain-Barre, severe peripheral or autonomic neuropathy, transverse myelitis, encephalitis, aseptic meningitis
  * Laboratory abnormality grade ≥3 for >7days (except nephritis grade 3-4, combined elevations of aspartate or alanine transaminase and total bilirubin, hyperglycemia, serum electrolytes/enzymes changes without clinical impact)
  * Febrile neutropenia, documented infection with absolute neutrophil count<10^9/L, grade 3 neutropenia >7days, grade 4 neutropenia or thrombocytopenia, or bleeding with platelet transfusion
  * AE with discontinuation >21days
  * Significant drug-related AE
Proportion of unacceptable toxicity of the regimen during the whole treatment course | 12 months or treatment discontinuation
  Presence of at least one of (composite endpoint):
  * Adverse event (AE) grade >3 (NCI-CTCAE v5), at least possibly related to the treatment or unrelated to disease, progression, intercurrent illness, concomitant medications
  * Non-hematological AE grade ≥3
  * Recurring grade 2 pneumonitis, Myocarditis grade ≥2
  * Autoimmune hemolytic anemia, hemolytic uremic syndrome, acquired hemophilia grade ≥3
  * Guillain-Barre, severe peripheral or autonomic neuropathy, transverse myelitis, encephalitis, aseptic meningitis
  * Laboratory abnormality grade ≥3 for >7days (except nephritis grade 3-4, combined elevations of aspartate or alanine transaminase and total bilirubin, hyperglycemia, serum electrolytes/enzymes changes without clinical impact)
  * Febrile neutropenia, documented infection with absolute neutrophil count<10^9/L, grade 3 neutropenia >7days, grade 4 neutropenia or thrombocytopenia, or bleeding with platelet transfusion
  * AE with discontinuation >21days
  * Significant drug-related AE
Proportion of patients with adverse events during the whole treatment course | 12 months or treatment discontinuation
  All adverse events during the whole treatment course
Duration of overall response | 24 months
  Time between the first occurrence of tumor objective response, partial or complete (RECIST 1.1) and the first radiological progression, with response assessment every 9 weeks, up to 24 months
Time to response | 24 months
  Time between inclusion and the first occurrence of tumor objective response (complete or partial, according to RECIST 1.1) or the end of the study, with response assessment every 9 weeks, up to 24 months
Progression-free survival | 24 months
  Time between inclusion and the date of the first radiological progression (according to RECIST 1.1), death (any cause), or last follow-up (maximum=24 months), whichever occurs first.
Overall survival | 24 months
  Time between inclusion and death (any cause) or last follow-up (maximum=24 months), whichever occurs first

CONTACTS AND LOCATIONS:
Locations (7):
- France (7):
  - Hôpital Jean Minjoz, Besançon
  - Centre François Leclerc, Dijon
  - Centre Léon Bérard, Lyon
  - AP-HP Hôpital Saint Louis, Paris
  - Hôpital Haut Lévêque, Pessac
  - Institut Universitaire du Cancer, Toulouse
  - Institut Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: Undecided